CLINICAL TRIAL: NCT01828437
Title: Addition of Pyridoxine to Prednisolone in the Treatment of Infantile Spasms: A Randomized Controlled Trial
Brief Title: Addition of Pyridoxine to Prednisolone in Infantile Spasms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Satinder Aneja, Director Professor and Head, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PYRIPREDIS
Record Dates: First submitted 2013-04-07; First posted 2013-04-10 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Infantile Spasms
MeSH Terms: conditions — Spasms, Infantile | interventions — Pyridoxine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pyridoxine plus prednisolone (Experimental): allocated patients receive pyridoxine (30 mg/kg/day) in addition to prednisolone
  Interventions: Drug: Pyridoxine plus prednisolone
- Prednisolone (Active Comparator): allocated patients receive prednisolone alone
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Pyridoxine plus prednisolone
  Arms: Pyridoxine plus prednisolone
Drug: Prednisolone
  Arms: Prednisolone

SUMMARY:
Infantile spasms constitute a unique age specific epilepsy syndrome of infancy, characterized by epileptic spasms often accompanied by neurodevelopmental regression and an EEG finding of hypsarrhythmia. When all 3 components are present, the eponym "West syndrome" is commonly used. West syndrome is a catastrophic epileptic encephalopathy. It does not respond well to standard anti-epileptic drugs. Hormonal therapy is the mainstay in the treatment of infantile spasms. This includes adreno-cortico trophic hormone (ACTH) and oral steroids. Variable dose of prednisolone used in the treatment. Oral prednisolone used in usual dose (2mg/kg) has been shown to be less effective as compared to ACTH. High dose prednisolone (4mg/kg) has been used in the treatment of infantile spasms, which has been shown to be as effective as ACTH. Pyridoxine has been used as first line treatment in Japan, however there is paucity of data on the efficacy of combination of pyridoxine with hormonal therapy. There are no studies comparing add on pyridoxine with high prednisolone versus high dose prednisolone alone in the treatment of infantile spasms. Therefore the study has been planned to see whether the addition of pyridoxine with high dose prednisolone in the treatment of infantile spasms improves the efficacy in terms of spasm cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Age in 3months-3years.
2. Presence of epileptic spasms (1 or more clusters per day) with EEG evidence of hypsarrythmia or its variants.

   -

Exclusion Criteria:

1. Children with active systemic illness
2. Children with evidence of active tuberculosis
3. Severe Acute Malnutrition (standard deviation scores below median weight for height)
4. Children with recurrent illness/chronic systemic illness
5. Prior treatment of pyridoxine, steroid, or ACTH.

   -

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children who achieved complete cessation spasm for at least 48 hours as per parental reports at the end of 2 weeks in both the groups. | 2 weeks
  Proportion of children who achieved complete cessation spasm for at least 48 hours as per parental reports at the end of 2 weeks in both the groups.

SECONDARY OUTCOMES:
• Proportion of children who achieved more than 50 % reduction of clinical spasms as per parental reports at the end of 2 weeks | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Satinder Aneja, MD, Principal Investigator — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College, New Delhi, India

REFERENCES:
- [Derived] Kunnanayaka V, Jain P, Sharma S, Seth A, Aneja S. Addition of pyridoxine to prednisolone in the treatment of infantile spasms: A pilot, randomized controlled trial. Neurol India. 2018 Mar-Apr;66(2):385-390. doi: 10.4103/0028-3886.227281. PMID 29547159